CLINICAL TRIAL: NCT05421728
Title: Effectiveness of Engaging in Advance Care Planning Talks (ENACT) Group Visits in Primary Care for Older Adults With and Without Alzheimer's Disease
Acronym: ENACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-1978; R01AG066804 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Advance Care Planning; Primary Health Care
Keywords: Advance Care Planning; Group Medial Visit; Shared Medical Appointment

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants: ENACT Group Visit (Experimental): Participants will engage in two 2-hour group visits related to advance care planning, including printed advance care planning resources.
  Interventions: Behavioral: ENACT group visit
- Participants: Mailed Resources (Active Comparator): Participants will receive printed advance care planning resources by mail.
  Interventions: Behavioral: Mailed Resources
- Clinic Stakeholders (No Intervention): Clinic stakeholders providing care for participants enrolled in the "Participants: Enact Group Visits" arm. Demographics, and adverse event data will not be collected for this arm.
- Caregivers (No Intervention): Caregivers will be consented via postcard consent to facilitate patient participants' engagement in the trial and group visits. Outcome measure, demographics, and adverse event data will not be collected for this arm, however caregivers will assist participants in providing outcome measure data (responding to surveys, etc.)

INTERVENTIONS:
Behavioral: ENACT group visit — Participation in two 2 hour group visits about advance care planning.
  Arms: Participants: ENACT Group Visit
Behavioral: Mailed Resources — Participants will receive advance care planning resources in the mail with instructions to follow up with their primary care provider.
  Arms: Participants: Mailed Resources

SUMMARY:
The main goal of the ENACT (ENgaging in Advance Care planning Talks) Group Visit intervention is to integrate a patient-centered advance care planning process into primary care, ultimately helping patients to receive medical care that is aligned with their values. The ENACT Group Visit intervention involves two group discussions about advance care planning with 8-10 patients who meet for 2-hour sessions, one month apart, facilitated by a geriatrician and a social worker. This study will compare the ENACT Group Visit intervention to mailed advance care planning materials.

DETAILED DESCRIPTION:
This pilot feasibility randomized controlled study will determine the feasibility, acceptability and preliminary efficacy of the ENACT Group Visit intervention compared to a comparison arm.

The ENACT Group Visit intervention aims to engage patients in an interactive discussion of key ACP concepts and support patient-initiated ACP actions (i.e. choosing decision-maker(s), deciding on preferences during serious illness, discussing preferences with decision-makers and healthcare providers, and documenting advance directives). The group visits involve two 2-hour sessions, one month apart, facilitated by a geriatrician and a social worker. The ENACT Group Visit is based on an intervention manual that guides the structure, facilitator considerations, session format, and documentation and billing details. The discussions include sharing experiences related to ACP, considering values related to serious illness, choosing a surrogate decision-maker(s), flexibility in decision making, and having conversations with decision-makers and healthcare providers. The facilitators support an interactive discussion that promotes opportunities for patients to learn from others' experiences.

ELIGIBILITY:
Patient Participants:

Inclusion Criteria:

* 70 or older
* At least one clinic visit in past year
* No advanced care planning (ACP) document in electronic health record based on a clinic-level, population-based report
* Preferred language English for UCHealth clinics or preferred language English or Spanish for Denver Health clinic

Exclusion Criteria:

* Inability to demonstrate informed consent
* Does not have ready access to a telephone
* Inability to travel to clinic
* Moving out of area in 6 months
* Inability to participate in group visits due to hearing impairment as determined by clinic and/or study staff
* A household member (same address) is already enrolled

Caregivers

Inclusion Criteria:

* Age 18 and older
* Preferred language English for UCHealth clinics or preferred language English or Spanish for Denver Health clinic
* Patient with potential cognitive impairment consented to participate in study

Exclusion Criteria:

* Does not have ready access to a telephone
* Inability to travel to clinic
* Moving out of area in 6 months
* Inability to participate in group visits due to hearing impairment as determined by clinic and/or study staff

Clinic Stakeholders

Inclusion Criteria:

* Work as a multidisciplinary team member at a participating primary care clinic in the study
* English speaking as a preferred language
* Invited to participate in interviews or focus groups after the ENACT Group Visits intervention

Exclusion Criteria:

- Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with New Advanced Care Planning (ACP) documentation in their electronic health record at 6 Months | 6 months
  Number of Participants with New Advanced Care Planning (ACP) documentation in the electronic health record inclusive of advance directives (i.e., easy-to-read advance directive, medical durable power of attorney forms, living wills), and medical orders (POLST forms or CPR directives. If an advanced care planning document is completed and in patient's electronic health record, the participant will be counted as having a New ACP.

SECONDARY OUTCOMES:
Measure of readiness for ACP | Baseline, 6 months
  Patient readiness for Advanced Care Planning (ACP) will be measured via the Advanced Care Planning (ACP) Engagement Survey. The 4-item ACP Engagement Survey assesses ACP readiness for signing papers for a decision maker; talking with a decision maker; talking with the doctor about future care; and signing papers about future care. Possible scores range from Possible scores for each item range from 1-5 and total scores range from 4-20, with higher indicating more planning readiness and a better outcome.
Measure of decision self-efficacy | Baseline, 6 months
  The 11-item Decision Self-Efficacy Scale measures self-confidence or belief in one's abilities in decision making. Possible scores range from 0 to 100, with higher scores indicating more decision self-efficacy and a better outcome.
The Quality of Communication (QOC) | Baseline, 6 months
  Quality of Communication (QOC) Questionnaire is a 13-item validated measure of the overall quality of end-of-life communication. Possible scores are averaged and range from 0 to 10, with higher scores indicating a better outcome.
Composite of advanced care planning documentation | Baseline, 6 months
  Clinician documentation of ACP (preferences for future medical care) in electronic health record will be measured using a standardized and double-adjudicated chart review audit process. The number of participants with clinician-documented ACP present in their electronic health records will be reported. Documentation of ACP that is added to the record as part of the ENACT group visits will be excluded.

OTHER OUTCOMES:
Percent of Recruitment (Reach) | From date of pre-screening until the date of participants' decision to enroll in study or not, up to 3 months
  Percent of individuals who participate of eligible patients, by clinic-based screening
Percent of Retention | 6 Months
  Percent of individuals who complete the intervention and the 6 month follow up
Telephone Montreal Cognitive Assessment (T-MoCA) scores | Baseline, 6 months
  The T-MoCA measures cognitive impairment in adults via a questionnaire conducted over the phone. Possible scores range from 0 to 22, with lower scores indicating a worse outcome.
Patient Reported Outcome Measurement Information System Global Health Scores | Baseline, 6 months
  The Patient Reported Outcomes Measurement Information System (PROMIS®) Global Health score measures patient reported measures of health. Scores are converted to a T score so that the average respondent score of 50 with a standard deviation of 10 points, with scores of higher than 50 indicating better than average outcomes, and scores of lower than 50 indicating worse than average outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Lum, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (8):
- United States (8):
  - UCHealth, Aurora, Colorado
  - UC Health Boulder Family Medicine, Boulder, Colorado
  - Denver Health Westside Clinic, Denver, Colorado
  - UC Health Lowry Internal Medicine, Denver, Colorado
  - UC Health AF Williams Family Medicine, Denver, Colorado
  - UC Health Lone Tree Seniors, Lone Tree, Colorado
  - UC Health Lone Tree Primary Care, Lonetree, Colorado
  - UC Health Westminster Primary Care, Westminster, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum HD, Jones J, Matlock DD, Glasgow RE, Lobo I, Levy CR, Schwartz RS, Sudore RL, Kutner JS. Advance Care Planning Meets Group Medical Visits: The Feasibility of Promoting Conversations. Ann Fam Med. 2016 Mar;14(2):125-32. doi: 10.1370/afm.1906. PMID 26951587
- [Derived] Farro SA, Juarez-Colunga E, Patel C, Bettcher BM, Haynes CA, Huebschmann AG, Nowels D, Tietbohl CK, Shi J, Ritger C, Shanbhag P, Resman K, Sudore RL, Lum HD. Engaging English- and Spanish-speaking older adults with and without possible cognitive impairment in advance care planning group visits: protocol for the ENgaging in Advance Care Planning Talks (ENACT) randomized controlled trial. Trials. 2025 Sep 25;26(1):353. doi: 10.1186/s13063-025-08964-x. PMID 40999430
- [Derived] Lum H, Farro S, Juarez-Colunga E, Patel C, Bettcher B, Haynes C, Huebschmann A, Nowels D, Tietbohl C, Shi J, Ritger C, Shanbhag P, Resman K, Sudore R. Engaging English- and Spanish-speaking older adults with and without possible cognitive impairment in advance care planning group visits: Protocol for the ENgaging in Advance Care Planning Talks (ENACT) Randomized Controlled Trial. Res Sq [Preprint]. 2025 Jun 20:rs.3.rs-6560971. doi: 10.21203/rs.3.rs-6560971/v1. PMID 40585266

DOCUMENTS (2):
  • Informed Consent Form: English Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT05421728/ICF_002.pdf
  • Informed Consent Form: Spanish Consent From (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT05421728/ICF_003.pdf